CLINICAL TRIAL: NCT04024865
Title: Use of Domperidone and Risk of Serious Cardiac Events in Postpartum Women
Brief Title: Domperidone and Risk of Serious Cardiac Events in Postpartum Women
Status: Completed | Type: Observational
Sponsor: Canadian Network for Observational Drug Effect Studies, CNODES (Other)
Collaborators: Drug Safety and Effectiveness Network, Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: Q16-10
Record Dates: First submitted 2019-07-12; First posted 2019-07-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2021-07

CONDITIONS: Ventricular Tachyarrhythmia; Sudden Cardiac Death; Lactation; Breast Feeding
Keywords: Domperidone; Postpartum; Ventricular Tachyarrhythmia; Sudden Cardiac Death
MeSH Terms: conditions — Tachycardia, Ventricular; Death, Sudden, Cardiac; Breast Feeding | interventions — Domperidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Treated with domperidone: Women who received a prescription for domperidone during the six months following delivery.
  Interventions: Drug: Domperidone
- Unexposed group (reference): Women with no prescription for domperidone during the six months following delivery.
  Interventions: Drug: No domperidone

INTERVENTIONS:
Drug: Domperidone — Women who received a prescription for domperidone (ATC A03FA03) during the six months following delivery.
  Other Names: ATC A03FA03
  Groups: Treated with domperidone
Drug: No domperidone — Women with no prescription for domperidone during the six months following delivery.
  Groups: Unexposed group (reference)

SUMMARY:
The purpose of this study is to determine whether the use of domperidone is associated with an increased risk of serious cardiac events among postpartum women in the six months following delivery. The hypothesis is that the use of domperidone will be associated with an increased risk of serious cardiac events among postpartum women.

The investigators will carry out separate population-based cohort studies using health care databases in five Canadian provinces. Women with live births will be eligible to enter the cohort. We will identify all women who start domperidone during the six months following delivery and match them to similar women who do not start domperidone, with all included women followed until the occurrence of an adverse cardiac event or for up to six months after delivery. The results from the separate sites will be combined to provide an overall assessment of the risk of serious cardiac events in users of domperidone.

DETAILED DESCRIPTION:
The overall objective of this study is to determine whether the use of domperidone is associated with an increased risk of serious cardiac events among postpartum women in the six months following delivery. More specifically, the investigators will assess whether domperidone is associated with the risk of ventricular tachyarrhythmia (VT) and sudden cardiac death (SCD).

A distributed, common-protocol approach will be used to conduct retrospective cohort studies using administrative health care data from five Canadian provinces (Alberta, British Columbia, Manitoba, Ontario and Saskatchewan). Briefly, the Canadian databases include population-level data on physician billing, diagnoses and procedures from hospital discharge abstracts, and dispensations for prescription drugs. The Ontario data will be restricted to social assistance recipients.

To assess this potential drug safety issue, the investigators will use a prevalent new-user cohort design as described by Suissa et al., 2017. In each jurisdiction, the investigators will first assemble a base cohort that includes all women aged between 15 and 55 years old with live births between April 1, 1997 and December 31, 2016 (or the latest available data at each site). Base cohort entry will be defined by the hospital discharge date after delivery. From this base cohort, a study cohort will be formed including all women who received a prescription for domperidone during the six months following delivery and matched women who have a physician visit at the same follow-up time and do not receive domperidone. Study cohort entry will be defined by the prescription date of domperidone for exposed women or the corresponding date of the physician visit for unexposed women. Women will be followed from the study cohort entry date until an event (defined below) or end of follow up (six months after delivery). Women will be permitted to contribute more than one observation to the study provided that each observation meets all the inclusion criteria.

Exposure to domperidone will be defined as a prescription for domperidone during the six months following delivery. Women not exposed to domperidone will serve as the reference group. Analyses will be conducted using an approach analogous to an intention-to-treat. Unexposed women who are subsequently exposed to domperidone will be censored at the time of the domperidone prescription. The primary outcome will be a composite endpoint of VT or SCD. Secondary outcomes will be the individual endpoints of VT, SCD, and all-cause mortality; separate follow-up durations will be estimated for each outcome.

Using a prevalent new-user design with time-based exposure sets, each user of domperidone will be matched to 10 unexposed women with a physician visit within ±30 days of the first domperidone dispensing of the exposed woman. Matching will be done on propensity score and calendar date of base cohort entry (i.e., hospital discharge from delivery hospitalization). Cox proportional hazards models will be used to estimate site-specific adjusted hazards ratios (HR) and corresponding 95% confidential intervals (CI) for each outcome of interest among postpartum women. Robust sandwich variance estimators will be used to account for potential within-subject clustering. As secondary analyses, the composite endpoint of VT or SCD will be stratified by domperidone dose and duration if feasible. Sensitivity analyses will be performed to assess the robustness of study results. Meta-analyses of the site-specific results will be performed using random-effects models.

In additional analyses, the demographic and clinical characteristics (including perinatal and peripartum characteristics) of women prescribed domperidone in the six months postpartum with those of women not prescribed it during this period will be compared. Furthermore, the impact of Health Canada safety advisories on prescribing patterns will be assessed via interrupted time series analyses.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 15 and 55 years old with live births between April 1, 1997 and December 31, 2016 (or the latest available data at each site)

Exclusion Criteria:

* Women with less than 365 days of healthcare coverage prior to the start of pregnancy
* Women with a domperidone prescription in the year prior to or during pregnancy
* Women with a diagnosis of Parkinson's disease or other diseases that cause autonomic dysfunction or use of antiparkinsonian agents anytime before delivery
* Women with a diagnosis of gastroparesis in the year prior to or during pregnancy
* Women with a diagnosis of ventricular tachyarrhythmia in the year prior to or during pregnancy

Ages: 15 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: In each jurisdiction, the investigators will assemble a base cohort that includes all women aged between 15 and 55 years old with live births between April 1, 1997 and December 31, 2016 (or the latest available data at each site). Base cohort entry will be defined by the hospital discharge date after delivery. From this base cohort, a study cohort will be formed including all women who received a prescription for domperidone during the six months following delivery and matched women who have a physician visit at the same follow-up time and do not receive domperidone. Study cohort entry will be defined by the prescription date of domperidone for exposed women or the corresponding date of the physician visit for the unexposed women.
Sampling Method: Probability Sample
Enrollment: 184929 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Ventricular tachyarrhythmia (VT) or sudden cardiac death (SCD) | Women will be followed from cohort entry until a diagnosis of VT or SCD, death, diagnosis of another indication for domperidone, end of healthcare coverage, or end of the study period (whichever occurs first), or for up to six months after delivery.
  VT or SCD will be identified with the following ICD codes:
  VT:
  ICD-9 codes 427.1, 427.4x; ICD-10 codes I47.0, I47.2, I49.0x
  SCD:
  ICD-9 codes: V12.53, 427.5, 798.1, 798.2, 798.9; ICD-10 codes: Z86.74, I46.x, R99, R96.0, R96.1, R98
  All potential SCD cases will be subjected to a computer algorithm to exclude non-relevant events (such as deaths occurring in hospital or due to non-cardiac pathology). At each site, computerized administrative records of potential SCD cases will be reviewed blinded to the exposure status to verify the accuracy of the algorithm. Finally, all potential cases that are not excluded by the algorithm will be manually reviewed in each site to ensure that all cases meet the event definition.

SECONDARY OUTCOMES:
All-cause mortality | Women will be followed from cohort entry until death from any cause, diagnosis of another indication for domperidone, end of healthcare coverage, or end of the study period (whichever occurs first), or for up to six months after delivery.
  All-cause mortality, which will include in-hospital and out-of-hospital death, will be defined by a recorded death in any database.

CONTACTS AND LOCATIONS:
Overall Officials: Kristian B Filion, PhD, Principal Investigator — McGill University
Locations (1):
- Lady Davis Institute for Medical Research, Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suissa S, Moodie EE, Dell'Aniello S. Prevalent new-user cohort designs for comparative drug effect studies by time-conditional propensity scores. Pharmacoepidemiol Drug Saf. 2017 Apr;26(4):459-468. doi: 10.1002/pds.4107. Epub 2016 Sep 9. PMID 27610604
- [Background] Moriello C, Paterson JM, Reynier P, Dahl M, Aibibula W, Fisher A, Gamble JM, Kuo IF, Ronksley PE, Winquist B, Filion KB; Canadian Network for Observational Drug Effect Studies (CNODES) Investigators. Off-label postpartum use of domperidone in Canada: a multidatabase cohort study. CMAJ Open. 2021 May 14;9(2):E500-E509. doi: 10.9778/cmajo.20200084. Print 2021 Apr-Jun. PMID 33990364
- See also: This is the organization's website describing general functions, other CNODES projects, and investigator profiles. — http://www.cnodes.ca